CLINICAL TRIAL: NCT02328222
Title: PHASE 4, STUDY OF THE EFFECT OF EARLY STEROID WITHDRAWAL IN RENAL TRANSPLANT RECEPIENTS OF A LIVING-RELATED DONOR
Brief Title: ESTEROID WITHDRAWAL STUDY, SAFETY AND EFFICACY IN RENAL TRANPLANTATION
Acronym: ESWMEX001
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Unidad de Investigacion Medica en Enfermedades Renales (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SWKT
Record Dates: First submitted 2014-07-15; First posted 2014-12-31 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2014-12

CONDITIONS: END STAGE RENAL DISEASE
Keywords: Early steroid withdrawal; Acute allograft rejection; Mycophenolate; Tacrolimus; Basiliximab
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CONTROL GROUP (No Intervention): CORTICOSTEDORID TREATMENT WAS AS FOLLOWS: day zero post-transplantation (DP 0), 500 mg/day of MPD; (DP 1), 250 mg MPD; (DP 2), 125 mg MPD; (DP 3), 60 mg MPD; (DP 4), 30 mg MPD; and (DP 5), PREDNISONE AS DOSES 1 MG/KG (1 MONTH) AND A REDUCTION TO ACHIEVE 0.1 MG/KG IN THE 3rd MONTH.
- ESW group (Experimental): CORTICOSTEDORID TREATMENT WAS AS FOLLOWS: day zero post-transplantation (DP 0), 500 mg/day of MPD; (DP 1), 250 mg MPD; (DP 2), 125 mg MPD; (DP 3), 60 mg MPD; (DP 4), 30 mg MPD; and (DP 5), PREDNISONE AS DOSES 1 MG/KG (1 MONTH) AND A REDUCTION TO ACHIEVE 0.1 MG/KG IN THE 3rd MONTH.
  Interventions: Drug: ESW group

INTERVENTIONS:
Drug: ESW group — CORTICOSTEDORID TREATMENT WAS AS FOLLOWS: day zero post-transplantation (DP 0), 500 mg/day of MPD; (DP 1), 250 mg MPD; (DP 2), 125 mg MPD; (DP 3), 60 mg MPD; (DP 4), 30 mg MPD; and (DP 5), PREDNISONE AS DOSES 1 MG/KG (1 MONTH) AND A REDUCTION TO ACHIEVE 0.1 MG/KG IN THE 3rd MONTH.
  Other Names: STEROID AVOIDANCE; STEROID WITHDRAWAL
  Arms: ESW group

SUMMARY:
BACKGROUND: Non-steroid maintenance immunosuppression after transplantation can improve long-term lipid and hemodynamic profiles without severe acute rejection (AR) events that alter graft function or survival. Our objective was to evaluate the effects of early steroid withdrawal (ESW) on the frequency and severity of AR using an immunosuppressive scheme consisting of mycophenolate (MMF) and tacrolimus (TAC) in combination with an induction treatment with basiliximab.

METHODS: A randomized clinical trial was performed on first renal transplant recipients. In the ESW group, patients were selected for corticosteroid treatment withdrawal on the fifth day post-transplantation. In the Control group, patients continued steroid treatment.

DETAILED DESCRIPTION:
INTRODUCTION New immunosuppressant drugs have lowered early acute rejection (AR) rates with controversial results on improved long-term renal graft and patient survival (1-3).

An ideal maintenance immunosuppressant treatment for an improved long-term renal graft function and survival has not been determined (4). With new and more potent immunosuppressants available, new strategies are being developed to reduce or eliminate the use of steroids after transplantation due to important side effects and the lack of benefit in long-term graft and patient survival (5-8).

Immunosuppression minimization strategies have led to the possibility of early steroid withdrawal with similar results for AR incidence, function, and renal graft as well as patient survival among those that continue steroid treatment after transplantation (9-21).

Current clinical practice guidelines for kidney disease improving global outcomes (KDIGO) suggest that steroids could be withdrawn from patients with low immunological risk after kidney transplantation when receiving induction immunosuppressive therapy (22). However, a recent meta-analysis indicated that steroid removal or withdrawal after renal transplantation could be linked to the risk of kidney graft AR on all immunosuppression regimens (5). Nevertheless, kidney graft rejection with non-steroidal immunosuppression shows mild rejection characteristics with no negative impact on function or graft and patient survival, but this type of intervention is still controversial (5).

In Mexico, there is no information concerning therapeutic intervention of steroid withdrawal after transplantation, and it is not common practice.

In our hospital, the highest percentage of kidney transplants consist of living-related donors with low immunological risk, in most cases on a steroid based-immunosuppressive regimen with mycophenolate mofetil (MMF) and calcineurin inhibitors; Tacrolimus (TAC) or cyclosporine (CsA) are used for maintenance immunosuppressive therapy (23). We believe that steroid withdrawal after transplantation could be beneficial due to the low immunological risk and the high risks of diabetes, obesity, and metabolic syndrome in our population (24, 25). Thus, the objective of this study was to assess and compare the effects of early steroid withdrawal on the frequency and severity of AR and its impact on function and graft survival.

MATERIALS AND METHODS The study was performed in the Division of Transplantation of the Specialties Hospital, Western National Medical Center, IMSS Guadalajara, Jalisco following the ethical norms of the Helsinki Declaration with approval of the local ethics committee and with written informed consent.

STUDY DESIGN A randomized, open-label, controlled clinical trial on patients that had a single kidney transplant using a living donor (related or non-related) was performed from June 2010 to June 2011. The patients underwent immunosuppressive maintenance treatments either without prednisone (PDN) (Early steroid withdrawal group) or with PDN (Control group). All patients were over 18 years of age with panel reactive antibody (PRA) class I and II HLA <20%. We excluded patients with co-morbidities that required the use of steroid, delayed graft function or AR during the 5 days post-transplantation, along with patients that decided to leave the study.

Variables such as ages and genders of the recipient and the donor, family history of diabetes mellitus, pregnancy, weight, height, blood pressure, glucose levels, lipid profile, cause of renal disease, HLA histocompatibility, PRA, cytomegalovirus (CMV) serostatus, and drug treatment (anti-hypertensive agents, euglycemic agents, statins) were obtained, as were the dates of diagnosis of dyslipidemia, high systemic blood pressure, or post-transplantation diabetes mellitus (PTDM). Posttransplant assessments were made at 3, 6, 9, and 12 months. Information collected included the date of the transplant, type of donor, cold and warm ischemic times, immunosuppressant-induction (basiliximab) and maintenance (TAC, MMF, PDN), date of AR diagnosis, and the anti-rejection treatment (methylprednisolone or thymoglobulin). The number of AR events, their severity, and the presence of chronic graft nephropathy were defined using the Banff classification (26).

The histopathological analysis of the graft was evaluated using protocolized percutaneous kidney biopsies at 3, 6, and 12 months post-transplantation. These biopsies were performed on patients that clinically required them, and the same pathologist analyzed the samples. The AR episodes (subclinical, borderline, and Banff 1A)(26) were managed with IV methylprednisolone (MPD), 250 mg to 1 g for 3 to 5 days, and with polyclonal antibodies (thymoglobulin) for steroid-resistant AR or severe AR (26) at a dose of 1.5 mg/kg/day for 7 to 10 days. In cases of humoral rejection, plasmapheresis and 300 mg/m2 of rituximab were considered.

Patients subjected to the protocol or those requiring biopsies and presenting histopathological evidence of borderline changes or IA-Banff classification were treated with MPD and continued in the study. Patients with severe AR or steroid-resistant AR were excluded from the study (but not the analysis), and steroid treatment was restarted after the AR event.

Renal function was determined with the following method: MDRD-4 formula (MDRD (ml/min/1.73 m2) = 186 x (creatinine /88.4)-1.154 x age-0.203 x 0.742 if female) (27).

TAC blood levels were measured via quantitative colorimetric analysis using a blood EMIT (enzyme-multiplied immunoassay technique) 2000 Tacrolimus Assay (Syva-SIEMENS). TAC levels in the first 30 days were maintained between 9-15 ng / ml, and from day 31 to 365, levels of 8-10 ng / ml were considered appropriate.

Class I and II HLA PRAs were determined before transplantation using Flow-PRA (One Lambda Inc, Canoga Park, CA, USA); a cut-off level of >20% was considered positive.

DEFINITIONS Early steroid withdrawal (ESW) is defined arbitrarily as the absence of steroids after the fifth day post-transplantation.

Post-transplantation diabetes mellitus (PTDM) is a hyperglycemic state posterior to transplantation occurring with fasting glucose of >126 mg/dl on two different occasions or a fasting random glucose of 200 mg/dl (28).

Systemic arterial hypertension (SAH) is when the blood pressure exceeds 140/90 mmHg, based on two or more measurements on two or more visits (29).

IMMUNOSUPPRESSION PROTOCOLS The immunosuppressive-induction scheme used on this study was based on 0.18 mg/kg/day of TAC in two doses, 2 g/day of mycophenolate mofetil (MMF) per day in two doses, 500 mg methylprednisolone before surgery (day zero), and anti-interleukin 2 humanized monoclonal antibodies (20 mg of basiliximab (Simulect®) on the first and fourth days post-transplantation. Maintenance immunosuppression was based on 2 g/day of MMF in two doses and 0.1-0.2 mg/kg/day of TAC in two doses (the doses were modified according to serum levels). Early steroid withdrawal was performed as follows: day zero post-transplantation (DP 0), 500 mg/day of MPD; (DP 1), 250 mg MPD; (DP 2), 125 mg MPD; (DP 3), 60 mg MPD; (DP 4), 30 mg MPD; and (DP 5), steroid suspension.

STATISTICAL ANALYSIS Continuous variables were analyzed using Student's t-test, and demographic categorical variables and result differences between the groups were analyzed using the chi-square test. To estimate the risk of rejection on steroid-withdrawal patients, a logistic regression analysis was performed. Rejection-free and graft survival were estimated using the Kaplan-Meier survival analysis. Results were considered significant with p<0.05. Statistical analysis was performed using the SPSS Statistical Package version 17.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Panel reactive antibody (PRA) class I and II HLA <20%.
* Any gender
* Living donor

Exclusion Criteria:

* Patients with co-morbidities that required the use of steroid,
* Delayed graft function or AR during the 5 days post-transplantation,
* Along with patients that decided to leave the study.
* Multiorganic recipients

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2010-06; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
ACUTE REJECTION FREQUENCY AND SEVERITY | UP TO 1 YEAR OF FOLLOW UP
  ACUTE REJECTION ACCORDING TO BANFF´S CLASSIFICATION, LIMITROPHIC CHANGES (1), ACUTE REJECTION 1A (2), 1B (3), 2A (4), 2B (5); CHRONIC REJECTION (6)

SECONDARY OUTCOMES:
RENAL GRAFT FUNCTION | UP TO 1 YEAR OF FOLLOW UP
  GRAFT FUNCTION IS MEASURED BY eGFR USING MDRD-4 FORMULAE, RESULTS ARE SHOWN IN ML/MIN

CONTACTS AND LOCATIONS:
Overall Officials: ALFONSO M CUETO-MANZANO, PhD, Study Director — Instituto Mexicano del Seguro Social
Locations (1):
- Umae Hospital de Especialidades, Guadalajara, Jalisco, Mexico